CLINICAL TRIAL: NCT06976671
Title: A Phase II Proof-of-concept Study Evaluating the Safety and Efficacy of Bevacizumab in the Treatment of Adhesive Capsulitis
Brief Title: A Study to Determine the Safety and Efficacy of Bevacizumab Administered Via Injection Into the Shoulder Joint of Participants With Adhesive Capsulitis (Frozen Shoulder)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MQ-SR-001
Record Dates: First submitted 2024-09-10; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-09

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis; Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: Participants will receive a single intra-articular dose of 50mg bevacizumab. This dose will increase sequentially by 50mg per treatment cohort, until otherwise stopped due to dose-limiting toxicities or Sponsor discretion.
  The dose-ranging follows a classic "3+3 design" to establish dose-limiting toxicities and the recommended dose for future studies. All dose escalations will be determined after a safety evaluation of the prior cohort. The design will be conducted as follows: initially, three participants will be enrolled into cohort 1 and will receive a 50mg dose of bevacizumab. The occurrence of a single treatment-related dose limiting toxicity will prompt enrolment of three additional participants into the same cohort. When more than one treatment-related dose limiting toxicity occurs in ≤ 6 patients in a dosing cohort, dose escalation will be stopped, and this dose level will be identified as the non-tolerated dose. Otherwise, if ≤ 1 treatment-related dose limiting toxicity occur
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intra-articular Bevacizumab (Experimental): Bevacizumab administered as a single-dose intra-articular injection at 4 dose levels (50mg, 100mg, 150mg, 200mg)
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — intra-articular bevacizumab

SUMMARY:
This study is intended to test a new treatment for a condition called adhesive capsulitis, also known as frozen shoulder. The treatment being tested is called bevacizumab. Participants will receive a single dose of bevacizumab (50mg, 100mg, 150mg, or 200mg) via injection into their shoulder joint. After the injection, participants will return to site 6 times over the course of a year for safety assessments, questionnaires to track pain levels, and range of movement tests conducted by a physiotherapist.

The main goal of this study is to:

1. Evaluate the safety and effectiveness of bevacizumab when it is injected into the frozen shoulder joint.
2. Determine the maximum dose of bevacizumab that can be given without side effects.

This is an investigator initiated clinical trial sponsored by Macquarie University. There will be a maximum of 28 participants enrolled and the only site involved in recruitment is Macquarie University.

DETAILED DESCRIPTION:
This study is a single-centred, open-label, dose-ranging clinical trial to assess the safety and efficacy of intra-articular bevacizumab in adults with adhesive capsulitis. Participants, aged 18 years and over, will be included in this study if they are diagnosed with adhesive capsulitis as defined in the inclusion criteria. Eligibility will be dependent on the exclusion of any previous shoulder trauma in the contralateral shoulder, previous adhesive capsulitis or any other differential diagnosis of the ipsilateral shoulder, and serology confirming absence of diabetes mellitus.

The dose-ranging follows a classic "3+3 design" to establish dose-limiting toxicities and the recommended dose for future studies. All dose escalations will be determined after a safety evaluation of the prior cohort. The design will be conducted as follows: initially, three participants will be enrolled into cohort 1 and will receive a 50mg dose of bevacizumab. The occurrence of a single treatment-related dose limiting toxicity (defined as a grade 3 or higher adverse event as per Common Terminology Criteria for Adverse Events version 5.0 [United States of Health and Human Services, 2017]) will prompt enrolment of three additional participants into the same cohort. When more than one treatment-related dose limiting toxicity occurs in ≤ 6 patients in a dosing cohort, dose escalation will be stopped, and this dose level will be identified as the non-tolerated dose. Otherwise, if ≤ 1 treatment-related dose limiting toxicity occurs in ≤ 6 participants, three participants will be enrolled into the next cohort (cohort 2) and receive a sequentially higher dose of bevacizumab (100mg). This will continue at 50mg increases of bevacizumab for each cohort unless otherwise stopped due to dose-limiting toxicities or Sponsor discretion. The maximum planned dose will be cohort 4 (200mg dose). For this cohort, it is planned to enroll up to 10 participants unless DLTs are observed or enrolment is stopped.

ELIGIBILITY:
Inclusion Criteria:

IC1. Over 18 years of age (inclusive) at the time of signing informed consent

IC2. Clinical diagnosis of adhesive capsulitis which is defined as:

1. Progressive pain and stiffness for a period greater than 2 months but less than 6 months; and,
2. Either thickening or signal hyperintensity associated with coracohumeral ligament, axillary pouch, or rotator interval joint capsule OR obliteration of the subcoracoid fat triangle as confirmed by radiological examination (magnetic resonance imaging); and,
3. Normal x-ray of the shoulder with no evidence of glenohumeral joint degenerative changes or sequelae of previous trauma.

IC3. Capable of giving signed informed consent as described in Section 14 of the protocol which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol

IC4. Participants of child-bearing potential are eligible to participate if they agree to the following during the study intervention period and for a minimum of 120 days after the study intervention is administered:

1. Female participants must not be pregnant or breastfeeding AND are either abstinent from heterosexual intercourse as their preferred usual lifestyle OR engage in an adequate method of contraception (i.e., the oral contraceptive pill, intrauterine device, or other)
2. Male participants must refrain from donating sperm AND are either abstinent from heterosexual intercourse as their preferred usual lifestyle OR must agree to use an adequate method of contraception/barrier method (i.e. condom and/or heterosexual partner engaging in an adequate method of contraception as previously described)

IC5. Participants who are not of child-bearing potential, defined as at least one or more of the following criteria, are eligible to participate in the study

1. Female participants in a post-menopausal state (defined as not experiencing menses for 12 consecutive months without an alternative cause)
2. Documented permanent sterilisation method (including, but not limited to, hysterectomy, bilateral salpingectomy, bilateral oophorectomy, and vasectomy)

Exclusion Criteria:

EC1. History of previous surgery or treatment with corticosteroid prior to screening, platelet-rich plasma, or anti-VEGF injections in the ipsilateral shoulder

EC2. History of adhesive capsulitis in ipsilateral shoulder

EC3. Presence of trauma in the affected shoulder unrelated to adhesive capsulitis

EC4 Advanced imaging features associated with calcific tendinopathy

EC5. Presence of uncontrolled hypertension (defined as systolic pressure > 140mmHg and diastolic pressure > 100mmHg)

EC6. Any medical history of cardiovascular disease, uncontrolled ischemic heart disease, acute myocardial infarction within 12 months of study entry, or any history of intracranial hemorrhage, stroke or a transient ischaemic attacks at any time

EC7. Presence of inflammatory arthritis (such as but not limited to: systemic lupus erythematosus, rheumatoid arthritis, reactive arthritis, etc.), Parkinson's disease, brain injury, osteoarthritis, bony glenohumeral pathology, hypothyroidism, neuromuscular disorders, or pre-diabetes or diabetes mellitus (defined by fasting glucose ≥7mmol/L and Hba1c ≥ 5.7%)

EC8. Participants currently taking corticosteroids, monoclonal antibody therapy, or other immunosuppressants which are deemed to impact the study endpoints

EC9. Planning to or have received treatment for the affected shoulder at any time during the study or prior to the study included but not limited to:

1. Intra-articular or intrabursal injection(s) of lidocaine, suprascapular nerve blocks; corticosteroids, electroanalgesic and/or thermoanalgesic modalities
2. Intra-articular or intrabursal injection(s) of sodium hyaluronate and/or glenohumeral distension arthrography
3. Surgical intervention

EC10. Progressive pain and stiffness in the affected shoulder that is for a period less than 2 months or greater than 6 months

EC11. Hypersensitivity to the study intervention, including any constituents thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study

EC12. Any active malignancy under treatment

EC13. Women who are pregnant and/or breastfeeding, or who plan to be pregnant in the following six months after study intervention

EC14. Participants not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions that might affect their safety or ability to complete the protocol or that may confound the efficacy or safety results of the trial

EC15. Participants are employees of the clinical study site or other individuals directly involved in the conduct of the study, or immediate family members of such individuals (in conjunction with Section 1.61 of the ICH-GCP Ordinance E6)

EC16. Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalised

EC17. Participants unable to provide written informed consent

EC18. Participants who have participated in other clinical trial within 1 month, have participated in another study within 6 months from the date of selection, or have planned for participation in another trial during the follow up period of this trial which is deemed by the Investigator to impact the planned study endpoints of this study

EC19. Acute illness within the 30 days prior to V1 that, in the opinion of the Investigator, affects the participant's ability to participate in the study.

EC20. Participants currently taking warfarin or any other anti-coagulation therapies.

EC21.Participants deemed with any condition which would preclude their use for study-related magnetic resonance imaging procedures, including but not limited to: morbid obesity, severe claustrophobia, and/or permanent pacemaker).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of bevacizumab over a 52-week period in participants with adhesive capsulitis | 52 Weeks
  * Incidence of adverse events (including medically significant changes in physical assessments, laboratory assessments, vital signs, and electrocardiogram), and serious adverse events, at 7 days (V3), 14 days (V4), 28 days (V5), 84 days (V6), 168 days (V7), and 364 days (V8)
  * Incidence of adverse events and serious adverse events at 3 days (V2)
Determine the maximum tolerated dose of intra-articular bevacizumab at 1 week (V3) per cohort | From start of treatment to 1 week after treatment
  Maximum tolerated dose as defined as the highest dose where 0 out of 3 participants or no more than 1 out of 6 participants experienced any dose-limiting toxicity (defined as a grade 3 or higher adverse event as per Common Terminology Criteria for Adverse Events version 5.0

SECONDARY OUTCOMES:
Evaluate the efficacy of bevacizumab over a 52-week period in participants with adhesive capsulitis | 52 weeks
  Change in passive global range of motion loss against contralateral shoulder at baseline (V1) versus 14 days (V4), 28 days (V5), 84 days (V6), 168 days (V7), and 364 days (V8)
Evaluate the efficacy of bevacizumab over a 52-week period in participants with adhesive capsulitis | 52 weeks
  Change in pain levels (assessed by a visual analogue scale: 0 to 100, higher score indicating worse outcome) at baseline (V1) versus 14 days (V4), 28 days (V5), 84 days (V6), 168 days (V7), and 364 days (V8).
Evaluate the efficacy of bevacizumab over a 52-week period in participants with adhesive capsulitis | 52 weeks
  Change in Shoulder Pain and Disability Index assessment (Roach, 1991) at baseline (V1) versus 14 days (V4), 28 days (V5), 84 days (V6), 168 days (V7), and 364 days (V8)
Evaluate the efficacy of bevacizumab over a 52-week period in participants with adhesive capsulitis | 52 weeks
  Change in Quick Disabilities of the Arm, Shoulder and Hand assessment (Work and Health, 2006) at baseline (V1) versus 14 days (V4), 28 days (V5), 84 days (V6), 168 days (V7), and 364 days (V8)
Evaluate the efficacy of bevacizumab over a 52-week period in participants with adhesive capsulitis | 52 weeks
  Categorical change in severity classification of global range of motion loss at baseline (V1) versus 14 days (V4), 28 days (V5), 84 days (V6), 168 days (V7), and 364 days (V8)

OTHER OUTCOMES:
Evaluate the safety of bevacizumab over a 52-week period in participants with adhesive capsulitis | 52 Weeks
  Incidence of study discontinuations and withdrawals due to adverse events at 3 days (V2), 7 days (V3), 14 days (V4), 28 days (V5), 84 days (V6), 168 days (V7), and 364 days (V8)
Evaluate the efficacy of bevacizumab over a 24-week period in participants with adhesive capsulitis | 24 weeks
  Change in passive global range of motion loss against contralateral shoulder at baseline (V1) versus 84 days (V6) and 168 days (V7)
Evaluate the efficacy of bevacizumab over a 24-week period in participants with adhesive capsulitis | 24 weeks
  Change in Shoulder Pain and Disability Index assessment (Roach, 1991) at baseline (V1) versus 84 days (V6) and 168 days (V7)
Evaluate the efficacy of bevacizumab over a 24-week period in participants with adhesive capsulitis | 24 weeks
  Change in Quick Disabilities of the Arm, Shoulder and Hand assessment (Work and Health, 2006) at baseline (V1) versus 84 days (V6) and 168 days (V7)
Evaluate the efficacy of bevacizumab over a 24-week period in participants with adhesive capsulitis | 24 weeks
  Categorical change in severity classification of global range of motion loss at baseline (V1) versus 84 days (V6) and 168 days (V7)

CONTACTS AND LOCATIONS:
Overall Officials: Sumit Raniga, BSC, MSC, MBCHB, FRACS, FAORTH, Principal Investigator — Macquarie Unniversity
Locations (1):
- Macquarie University, North Ryde, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided